CLINICAL TRIAL: NCT04283071
Title: The Evaluation of Upper Limb Function in Multiple Sclerosis Using Kinematic Assessment
Brief Title: Kinematic Assessment In Multiple Sclerosis
Acronym: KAIMS
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: NE19/126048
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis
Keywords: Upper limb function; Kinematic assessment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Progressive MS patients administered clinical examination measures including EDSS, nine-hole PEG test, patient reported outcomes measures and kinematic assessment of upper limb function
  Interventions: Device: Boxed infrared gross kinematic assessment tool
- Control: Healthy volunteers administered nine-hole PEG test and kinematic assessment of upper limb function
  Interventions: Device: Boxed infrared gross kinematic assessment tool

INTERVENTIONS:
Device: Boxed infrared gross kinematic assessment tool — An optical motion capture system, which records the movements of infrared emitting diodes (IREDs) in three-dimensional (3D) space by triangulating images from a pair of infrared cameras

SUMMARY:
Multiple sclerosis (MS) affects more than a 120,000 people in the United Kingdom and is the commonest neurological condition in young adults. MS causes a number of symptoms including weakness, altered sensation, pain and memory difficulties. There are different forms of MS, including relapsing-remitting MS (RRMS), primary progressive MS (PPMS) and secondary progressive MS (SPMS). Currently there are several effective treatments for RRMS, but no NICE approved treatment for SPMS. Patients with PPMS and SPMS experience a gradual progression in disability that affects individual patients differently. A number of clinical scores are used to quantify the disability in individual patients and some of these scores focus on the patients' lower limb function. In the progressive forms of MS, preservation of upper limb function becomes a more important concern for patients to maintain their quality of life.

With the advent of new treatment trials for PPMS and SPMS, it is important that clinicians and researchers are able to use accurate and quantifiable measures of upper limb function to evaluate any changes with time or response to treatment. The use of motion tracking software provides a unique opportunity to accurately track movements in real time and space and give a tailored assessment of an individual's function.

The overall aim of this study is to use established kinematic assessment tools to explore the extent and progression of upper limb dysfunction in patients with progressive MS. This aim will be achieved via the following objectives:

* Recruit a sample of participants with PPMS and SPMS from the local MS population
* Quantify the physical impairment in these participants using existing clinical scores as well the kinematic assessment tools that have been developed
* Follow-up the participants for a period of 12 months to identify and quantify any progression in their upper limb dysfunction
* Identify any factors that may influence upper limb dysfunction in this group
* Develop and evaluate the role of further kinematic techniques in this group of participants

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years at the time of enrolment into the study
* Participants with a confirmed diagnosis of MS that have entered the primary or secondary progressive stage for at least 12 months
* Participants must be able to comply with the terms and methods of the protocol
* Study specific written informed consent has been obtained

Exclusion Criteria:

* Age below 18 years at the time of enrolment into the study
* Participants with a diagnosis of RRMS
* Participants unable to comply with the terms or methods of the protocol
* Participants who report any cognitive or memory impairment
* Participants with significant co-morbidities that affect their upper limb function i.e. stroke etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or secondary progressive multiple sclerosis who report an impairement in their hand function
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in upper limb kinematic function in patients with progressive multiple sclerosis | 12 months
  Kinematic function will be measured using the Boxed Infrared Kinematic Assessment Tool

SECONDARY OUTCOMES:
Change in 9-hole PEG test performance in patients with progressive multiple sclerosis | 12 months
  The 9HPT is a brief, standardized, quantitative test of upper extremity function. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The two trials for each hand are averaged.
Change in EDSS in patients with progressive multiple sclerosis | 12 months
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time.
Change in patient reported outcome measures in patients with progressive multiple sclerosis | 12 months
  The ABILHAND and AMSQ-SF questionnaires will be administered to participants in the trial

OTHER OUTCOMES:
Association between upper limb kinematic function and 9-hole PEG test and EDSS in progressive multiple sclerosis | 12 months
  The kinematic measures used in this study will be compared to the use of current standard measures of testing function in multiple sclerosis, like the 9 hole PEG test and the EDSS

CONTACTS AND LOCATIONS:
Overall Officials: Linford Fernandes, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No